CLINICAL TRIAL: NCT00486239
Title: Emotional Processing and Memory Evaluation in Epilepsy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 08-06-06
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; memory; emotion
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Behavioral TLE 1A
  Interventions: Behavioral: TLE Arm 1; Behavioral: Emotion Memory Test
- 2 (Experimental): TLE Arm II
  Interventions: Behavioral: Emotion Memory Testing
- B (Experimental): Control Arm B
  Interventions: Behavioral: Emotion Memory Testing

INTERVENTIONS:
Behavioral: TLE Arm 1 — Behavioral/cognitive testing
  Arms: 1
Behavioral: Emotion Memory Test — Behavioral/cognitive Measure
  Arms: 1
Behavioral: Emotion Memory Testing — Behavioral/cognitive testing
  Arms: 2
Behavioral: Emotion Memory Testing — Behavioral/cognitive testing
  Arms: B

SUMMARY:
The purpose of the study is to assess the effects of temporal lobe epilepsy (TLE) on memory and emotional functioning. The study will evaluate the known lateralized neurological dysfunction(Right TLE versus Left TLE) on emotional verbal and visual memory function. Study data will assess the ability of participants with known lateralized neurological dysfunction (Right TLE versus Left TLE) to differentially perceive emotional stimuli. Another component of the study will evaluate possible changes in memory function for emotionally charged material following right or left temporal lobectomy for the treatment of medically intractable epilepsy. It is expected participants with known lateralized dysfunction will exhibit differential ability to discriminate emotional charged visual and verbal material.

DETAILED DESCRIPTION:
Epilepsy is a relatively common neurological disorder diagnosed when individuals suffer from repeated unprovoked seizures. Estimates of prevalence rates vary, but it is generally considered to be about 1% of the U.S. population. Of the patients diagnosed with epilepsy, about 60-70 percent are diagnosed with complex-partial seizures, and of these about 30-40 percent are medication refractory. The majority of individuals with medically refractory epilepsy have seizures arising from the temporal lobe area, labeled as Temporal Lobe Epilepsy (TLE). Patients with TLE experience neurological and psychiatric comorbidity. The surgical treatment of patients with medically refractory epilepsy has become increasingly recognized as an effective treatment to reduce or eliminate seizures in selected patients. Up to 90 percent of selected participants with TLE have been seizure free for a year following temporal lobectomy. However, patients undergoing neurological surgery for medication refractory epilepsy can experience a variety of cognitive and emotional comorbid complications. These include declines in memory and language functions as well as onset of depression, anxiety, and, rarely, de novo psychosis has been reported. This study will assess the material specific memory and emotion functioning of subjects with medically refractory temporal lobe epilepsy.

The incorporation of neuropsychological assessment in the pre-surgical evaluation of patients diagnosed with medically refractory epilepsy has been successful in reducing the risk of individuals experiencing catastrophic declines in memory and language functioning following neurological surgery. However, material specific memory loss remains a problematic issue in the surgical treatment for TLE. Despite 30 years of research, there remains questions about the lateralized function of mesial temporal structures. In addition, it has become increasingly recognized emotional function in patients with medically refractory epilepsy are related to quality of life and functional outcomes following temporal lobectomy. Indeed, post-surgical symptoms of depression and anxiety are significantly related to patient quality of life and, to a lesser extent, seizure freedom. Initial results suggested patients with right TLE were at greater risk for post-surgical emotional difficulties; however, more recent data question earlier observations and suggest hemisphere dominance has little affect on psychiatric outcome.

There is little doubt neurological surgery for medically refractory can significantly decrease, and in many instances, eliminate seizures in patients. However, individuals are at risk for cognitive and emotional comorbidity with these medical treatments and there remains a paucity of empirical study to help guide treatment. Despite increasing empirical evaluation of emotional (psychiatric) status in individuals with medically refractory epilepsy, there is a paucity of data exploring the interaction of learning and emotion functions. The purpose of this study is to prospectively evaluate the memory functioning of individuals with medically refractory TLE for emotional material. In addition, a component of the study will evaluate if there are differences in the ability to evaluate the emotional content of stimuli. Data from participants with epilepsy will be compared to a control group of healthy volunteers. The stimuli will consist of positive and negative material. It is suspected these data will, in the future, improve the pre-surgical evaluation of individuals with medically refractory epilepsy and reduce risk of the person having a pronounced psychiatric complication following temporal lobectomy.

ELIGIBILITY:
Inclusion Criteria:

* Referred to neurological institute at University Hospitals Case Medical Center for care of seizures/epilepsy
* Referred to neuropsychology laboratory for evaluation
* Participants must complete the routine check-in of all patients and sign consent and HIPAA forms.
* Be, in the investigator's opinion, compliant, able to follow the investigator's instructions and visit the clinic on schedule, cooperative and reliable.
* Be aged 18-64 years old.
* Be able to provide documented informed consent.
* Have a confirmed diagnosis of right or left temporal lobe epilepsy (TLE), which is made independent of their pre-surgical neuropsychological evaluation. Neurological disease must be confirmed by one (or more) of the following: (a) MRI study of the head, (b) CT study of the head, (c) EEG study, (d) Video-EEG study, (e) PET study of the head, (f) Neurological and Psychiatric exam by a physician.

Exclusion Criteria:

* Referred from an attorney or their evaluation is part of a personal injury claim.
* Be intoxicated from alcohol or other illicit substance.
* Received Electroconvulsive (ECT) treatment within the last 21 days.
* Have an MMSE score of 25 or less
* Have undergone Deep Brain Stimulator (DBS) surgery

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the effects of known lateralized neurological dysfunction (Right TLE versus Left TLE) on emotional memory function. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mike R Schoenberg, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States